CLINICAL TRIAL: NCT03162055
Title: A Randomised, Double-Blind, Double-Dummy, Multicentre, Parallel Group Study to Assess the Efficacy and Safety of Glycopyrronium/Formoterol Fumarate Fixed-dose Combination Relative to Umeclidinium/Vilanterol Fixed-dose Combination Over 24 Weeks in Patients With Moderate to Very Severe Chronic Obstructive Pulmonary Disease (AERISTO)
Brief Title: Efficacy and Safety of Glycopyrronium/Formoterol Fumarate Fixed-dose Combination Relative to Umeclidinium/Vilanterol Fixed-dose Combination Over 24 Weeks in Patients With Moderate to Very Severe Chronic Obstructive Pulmonary Disease
Acronym: AERISTO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel International Ltd (Unknown); Cognizant Technology Solution (Unknown); CISCRP (Industry); eResearchTechnology (Industry); QuintilesIMS Limited (Unknown); Corporate Translations Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D5970C00002
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Results first posted 2019-05-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-04

CONDITIONS: Chronic Obstructive Pulmonary Disease COPD
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate; Formoterol Fumarate; GSK573719; vilanterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): glycopyrronium/formoterol fumarate 7.2/4.8 μg per actuation, twice daily
  Interventions: Drug: Glycopyrronium/Formoterol Fumarate
- Active comparator (Active Comparator): umeclidinium/vilanterol 62.5/ 25μg per inhalation, once daily
  Interventions: Drug: umeclidinium/vilanterol

INTERVENTIONS:
Drug: Glycopyrronium/Formoterol Fumarate — Metered dose inhaler (MDI), contains glycopyrronium/formoterol fumarate fixed-dose combination 7.2/4.8 μg per actuation
  Arms: Experimental
Drug: umeclidinium/vilanterol — Dry powder inhaler (DPI), Each metered dose contains umeclidinium/vilanterol 62.5/ 25μg fixed-dose combination per inhalation
  Arms: Active comparator

SUMMARY:
This is a phase IIIb randomised, double-blind, double-dummy, multicentre, parallel group, 24 week study to assess the efficacy and safety of Glycopyrronium/Formoterol Fumarate (GFF) fixed-dose combination 7.2/4.8 μg 2 inhalations twice daily compared to Umeclidinium/Vilanterol (UV) 62.5/25 μg fixed-dose combination 1 inhalation once daily in Patients with moderate to very severe COPD.

ELIGIBILITY:
Inclusion criteria:

* Age 40-95 years at screening
* Current or former smoker with a history of at least 10 pack-years of cigarette smoking
* Current clinical diagnosis of COPD, with COPD symptoms > 1 year prior to screening, as defined by GOLD criteria or other current guidelines
* COPD Severity defined by FEV1/FVC ratio <0.70 and FEV1 <80% of predicted normal value at screening and at randomisation
* COPD treatment with rescue medication only, or stable dose of maintenance monotherapy (LAMA, LABA or ICS), or stable dose of double maintenance therapy (LAMA/LABA or ICS/LABA), for one month prior to screening
* COPD Assessment Test (CAT) score ≥10 at randomisation
* Documentation of a chest x-ray (as per local practice) or computed tomography (CT) within 6 months prior to screening, with no clinically significant pulmonary abnormalities other than related to COPD

Exclusion criteria:

* Respiratory disease other than COPD, including:
* Current diagnosis of asthma
* Alpha-1 Antitrypsin Deficiency as the cause of COPD
* Other respiratory disorders and conditions as listed in the protocol
* Severe COPD exacerbation (resulting in hospitalisation) not resolved within 8 weeks prior to screening, or moderate exacerbation not resolved within 4 weeks, or during screening
* Pneumonia or lower respiratory tract infection that required antibiotics within 8 weeks prior to screening, or during screening.
* Significant diseases or conditions other than COPD which may put the patient at risk, or influence the results of the study or the patient's ability to participate, including cardiac disease, advanced renal disease, and cancer that has not been in complete remission for at least 5 years.
* Patients who have needed additions or alterations to their usual maintenance therapy for COPD due to worsening symptoms within 1 month prior to and during screening
* Treatment with depot corticosteroids within 6 weeks, or other systemic corticosteroids within 4 weeks, prior to screening. (Patients maintained on an equivalent of 5 mg prednisone per day for at least 3 months prior to screening are allowed.)

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1119 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (84):
- United States (15):
  - Research Site, Tempe, Arizona
  - Research Site, Escondido, California
  - Research Site, Sacramento, California
  - Research Site, Hollywood, Florida
  - Research Site, Lawrenceville, Georgia
  - Research Site, Rincon, Georgia
  - Research Site, Farmington Hills, Michigan
  - Research Site, The Bronx, New York
  - Research Site, Gastonia, North Carolina
  - Research Site, Dublin, Ohio
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Greenville, South Carolina
  - Research Site, Spartanburg, South Carolina
  - Research Site, Sherman, Texas
  - Research Site, Tomball, Texas
- Bulgaria (15):
  - Research Site, Dupnitsa
  - Research Site, Haskovo
  - Research Site, Kozloduy
  - Research Site, Pazardzhik
  - Research Site, Petrich
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Razlog
  - Research Site, Rousse
  - Research Site, Sliven
  - Research Site, Smolyan
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
  - Research Site, Vidin
- Canada (10):
  - Research Site, Sherwood Park, Alberta
  - Research Site, Winnipeg, Manitoba
  - Research Site, Truro, Nova Scotia
  - Research Site, Burlington, Ontario
  - Research Site, Etobicoke, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Gatineau, Quebec
  - Research Site, Lévis, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
- France (8):
  - Research Site, Besançon
  - Research Site, Brest
  - Research Site, Lyon
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Pessac
  - Research Site, Poitiers
  - Research Site, Reims
- Hungary (13):
  - Research Site, Balassagyarmat
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Farkasgyepü
  - Research Site, Hajdúnánás
  - Research Site, Komárom
  - Research Site, Komló
  - Research Site, Miskolc
  - Research Site, Püspökladány
  - Research Site, Siófok
  - Research Site, Szeged
  - Research Site, Szombathely
  - Research Site, Vásárosnamény
- Russia (13):
  - Research Site, Barnaul
  - Research Site, Chelyabinsk
  - Research Site, Izhevsk
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Penza
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Saratov
  - Research Site, Smolensk
  - Research Site, Tomsk
  - Research Site, Ulyanovsk
  - Research Site, Yekaterinburg
- Ukraine (10):
  - Research Site, Chernivtsi
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Lutsk
  - Research Site, Lviv
  - Research Site, Odesa
  - Research Site, Poltava
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maltais F, Ferguson GT, Feldman GJ, Deslee G, Bourdin A, Fjallbrant H, Siwek-Posluszna A, Jenkins MA, Martin UJ. A Randomized, Double-Blind, Double-Dummy Study of Glycopyrrolate/Formoterol Fumarate Metered Dose Inhaler Relative to Umeclidinium/Vilanterol Dry Powder Inhaler in COPD. Adv Ther. 2019 Sep;36(9):2434-2449. doi: 10.1007/s12325-019-01015-3. Epub 2019 Jul 2. PMID 31267366

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 110 centers in 7 countries (Russia, Bulgaria, Ukraine, United States of America, Canada, Hungary and France) between 25 May 2017 and 04 May 2018. Participants with moderate to very severe chronic obstructive pulmonary disease (COPD) were recruited in this study.
Pre-assignment Details: The study had a screening period, followed by a 24-week double-blind and double-dummy treatment period. A total of 1445 participants were screened. Of which, 1119 participants were enrolled and randomized to study treatment.
Groups:
- Glycopyrronium/Formoterol Fumarate: Participants were randomized to receive 2 inhalations of glycopyrronium/formoterol fumarate (GFF) fixed-dose combination 7.2/4.8 micrograms (mcg) per actuation administered in the morning and evening by metered dose inhaler (MDI) for 24 weeks. Participants also received 1 inhalation of placebo matched to umeclidinium/vilanterol (UV) administered once daily in the morning by dry powder inhaler (DPI) for 24 weeks.
- Umeclidinium/Vilanterol: Participants were randomized to receive 1 inhalation of UV fixed-dose combination 62.5/25 mcg per actuation administered once daily in the morning by DPI for 24 weeks. Participants also received 2 inhalations of placebo matched to the GFF administered twice daily in the morning and evening by MDI for 24 weeks.
Period: Overall Study
Arm/Group | Glycopyrronium/Formoterol Fumarate | Umeclidinium/Vilanterol
Started | 559 | 560
Received Treatment | 557 | 560
Safety Analysis Set | 552 | 552
Full Analysis Set (FAS) | 552 | 552
Per Protocol (PP) Analysis Set | 506 | 510
Completed | 497 | 517
Not Completed | 62 | 43
Not completed — Adverse Event | 6 | 5
Not completed — Death | 3 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Study-specific withdrawal criteria | 22 | 14
Not completed — Withdrawal by Subject | 17 | 2
Not completed — Did not receive treatment | 2 | 0
Not completed — Incorrect randomization | 4 | 3
Not completed — Other | 8 | 15

BASELINE CHARACTERISTICS:
Population: The FAS included all randomized participants who received at least 1 inhalation of investigational product (IP) from the GFF or UV inhaler (active or placebo).
Groups:
- Glycopyrronium/Formoterol Fumarate: Participants were randomized to receive 2 inhalations of GFF fixed-dose combination 7.2/4.8 mcg per actuation administered in the morning and evening by MDI for 24 weeks. Participants also received 1 inhalation of placebo matched to UV administered once daily in the morning by DPI for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Glycopyrronium/Formoterol Fumarate | Umeclidinium/Vilanterol | Total
Number analyzed (Participants) | 552 | 552 | 1104
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.3 (8.0) | 63.8 (8.1) | 64.1 (8.0)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 273 | 292 | 565
  65 - 74 years | 223 | 214 | 437
  75 - 84 years | 53 | 43 | 96
  >=85 years | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 160 | 302
  Male | 410 | 392 | 802
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 10 | 23
  White | 538 | 542 | 1080
  More than one race | 0 | 0 | 0
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Morning Pre-dose Trough Forced Expiratory Volume in 1 Second (FEV1) Over 24 Weeks
Description: To assess the effects of GFF relative to UV on lung function as measured by change from baseline in morning pre-dose trough FEV1 is defined as the average of the -60 and -30 minute pre-dose values at each visit minus baseline using spirometry. Baseline is defined as the mean of the non-missing -60 and -30 minute values obtained prior to dosing at randomization (Day 1). BR a/s = bronchodilator responsiveness to albuterol/salbutamol.
Time Frame: From Baseline (Day 1) up to 24 weeks
Population: The PP analysis set included the subset of the FAS containing participants with post-randomization data obtained prior to important protocol deviations which may have affected efficacy. Only participants with data available for analysis are presented.
Measure: Least Squares Mean (Standard Error); unit: milliliter (mL)
Arm/Group | Glycopyrronium/Formoterol Fumarate | Umeclidinium/Vilanterol
Number analyzed (Participants) | 506 | 510
milliliter (mL) | 82.4 (11.2) | 169.6 (11.2)
Statistical Analysis 1: Comparison: Glycopyrronium/Formoterol Fumarate vs Umeclidinium/Vilanterol; Test type: Non-Inferiority — Non-inferiority p-value is calculated corresponding to the non-inferiority margin -50 mL; p = 0.9974, Repeated measures analysis; Change from baseline = Treatment + baseline FEV1 + BR a/s MDI + stratification factor (prior treatment) + region + visit + treatment by visit; Least Square Mean Difference = -87.2, 97.5% CI 2-sided [-117.0 to -57.4], Standard Error of Mean 13.3 — Estimate of the mean change from baseline over 24 weeks in the GFF treatment group is compared to the UV treatment group using a repeated measures analysis

2. Primary Outcome: Mean Peak Change From Baseline in FEV1 Within 2 Hours Post-dosing Over 24 Weeks in PP Analysis Set Population
Description: To assess the effects of GFF relative to UV on lung function in PP analysis set population as measured by peak change from baseline in FEV1 is defined as the maximum of the FEV1 assessments within the 2 hours post-dosing time windows at each visit minus baseline using spirometry. Baseline is defined as the mean of the non-missing -60 and -30 minute values obtained prior to dosing at randomization (Day 1).
Time Frame: From Baseline (Day 1) up to 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Glycopyrronium/Formoterol Fumarate | Umeclidinium/Vilanterol
Number analyzed (Participants) | 506 | 510
mL | 293.5 (10.2) | 296.9 (10.3)
Statistical Analysis 1: Comparison: Glycopyrronium/Formoterol Fumarate vs Umeclidinium/Vilanterol; Test type: Non-Inferiority — Non-inferiority p-value is calculated corresponding to the non-inferiority margin -50 mL; p = 0.0002, Repeated measures analysis; [statistical method as in outcome 1, analysis 1]; Least Square Mean Difference = -3.4, 97.5% CI 2-sided [-32.8 to 25.9], Standard Error of Mean 13.1 — Estimate of the mean peak change from baseline over 24 weeks in the GFF treatment group is compared to the UV treatment group using a repeated measures analysis

3. Secondary Outcome: Percentage of Participants With Increase of FEV1 of >=100 mL From Baseline at 5 Minutes Post-dosing on Day 1
Description: The percentage of participants with an increase in FEV1 of >=100 mL from baseline at 5 minutes post-dosing on Day 1 was determined to assess the early onset of action. Baseline is defined as the average of available evaluable -60 and -30 minute pre-dose assessments conducted at randomization (Day 1). Only data assigned to the 5 minute window was used to determine response. Participants with missing data were considered non-responders for the analysis.
Time Frame: 5 minutes post-dose on Day 1
Population: The FAS analysis set included all randomized participants who received at least 1 inhalation of IP from the GFF or UV inhaler (active or placebo).
Measure: Number; unit: Percentage of participants
Arm/Group | Glycopyrronium/Formoterol Fumarate | Umeclidinium/Vilanterol
Number analyzed (Participants) | 552 | 552
Percentage of participants | 60.1 | 40.8
Statistical Analysis 1: Comparison: Glycopyrronium/Formoterol Fumarate vs Umeclidinium/Vilanterol; Test type: Superiority; p < 0.0001, Regression, Logistic; ln (1/(1-p))=Treatment+baseline FEV1+BR a/s MDI+stratification factor (prior treatment)+region.p=percentage of participants with increase of >=100 mL; Odds Ratio (OR) = 2.30, 95% CI 2-sided [1.79 to 2.95] — Estimate of the log odds of being a responder in the GFF treatment group compared to the UV treatment group using a logistic regression

4. Secondary Outcome: Mean Peak Change From Baseline in Inspiratory Capacity (IC) Within 2 Hours Post-dosing Over 24 Weeks
Description: Peak change from baseline in IC is defined as the maximum of the IC assessments within the 2 hours post-dosing time windows at each visit minus baseline. Baseline is defined as the average of available evaluable -60 and -30 minute pre-dose assessments conducted at randomization (Day 1).
Time Frame: From Baseline (Day 1) up to 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Glycopyrronium/Formoterol Fumarate | Umeclidinium/Vilanterol
Number analyzed (Participants) | 506 | 510
mL | 363.1 (15.5) | 378.3 (15.6)
Statistical Analysis 1: Comparison: Glycopyrronium/Formoterol Fumarate vs Umeclidinium/Vilanterol; Test type: Non-Inferiority — Non-inferiority p-value is calculated corresponding to the non-inferiority margin -50 mL; p = 0.0371, Repeated measures analysis; Change from baseline = Treatment + baseline IC + BR a/s MDI + stratification factor (prior treatment) + region + visit + treatment by visit; Least Square Mean Difference = -15.2, 95% CI 2-sided [-53.4 to 22.9], Standard Error of Mean 19.4 — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Mean Transition Dyspnea Index (TDI) Focal Score Over 24 Weeks
Description: The baseline dyspnea index (BDI) and TDI consist of 3 individual components: functional impairment, magnitude of task, and magnitude of effort. For the BDI, each of these 3 components were rated in 5 grades from 0 (very severe) to 4 (no impairment), and were summed to form a baseline total score from 0 to 12. For the TDI, changes in dyspnea were rated for each component by 7 grades from -3 (major deterioration) to +3 (major improvement), and were added to form a TDI focal score from -9 to +9. Baseline is defined as the latest BDI assessment within 7 days before or at randomization (Day 1).
Time Frame: From Baseline (Day -7 or 1) up to 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Glycopyrronium/Formoterol Fumarate | Umeclidinium/Vilanterol
Number analyzed (Participants) | 506 | 510
Units on a scale | 1.23 (0.10) | 1.60 (0.10)
Statistical Analysis 1: Comparison: Glycopyrronium/Formoterol Fumarate vs Umeclidinium/Vilanterol; Test type: Non-Inferiority — Non-inferiority p-value is calculated corresponding to the non-inferiority margin -1.0 unit; p < 0.0001, Repeated measures analysis; TDI focal score = Treatment + Baseline Dyspnea Index + BR a/s MDI + stratification factor (prior treatment) + region + visit + treatment by visit; Least Square Mean Difference = -0.37, 95% CI 2-sided [-0.59 to -0.14], Standard Error of Mean 0.12 — Estimate of the mean TDI focal score over 24 weeks in the GFF treatment group is compared to the UV treatment group using a repeated measures analysis

6. Secondary Outcome: Mean Change From Baseline in Early Morning Symptoms of COPD Instrument (EMSCI) Over 24 Weeks
Description: Change from baseline in the 6-item EMSCI Symptom Severity Score was derived by averaging the responses from a participant on the 6 item-level symptom scores (scored on a 4-point scale from 1 to 4, whereas 1= mild and 4= very severe). The EMSCI collected data about the frequency and severity of early morning symptoms and the impact of COPD symptoms on early morning activity in participants with COPD. Participants completed a daily electronic patient-reported outcome (ePRO) questionnaire for their COPD symptoms. Baseline is defined as the average of the non-missing values from the ePRO data collected in the last 7 days before the randomization (Day 1). TI = Time interval.
Time Frame: From Baseline (Day -7) up to 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Glycopyrronium/Formoterol Fumarate | Umeclidinium/Vilanterol
Number analyzed (Participants) | 506 | 510
Units on a scale | -0.142 (0.018) | -0.176 (0.018)
Statistical Analysis 1: Comparison: Glycopyrronium/Formoterol Fumarate vs Umeclidinium/Vilanterol; Test type: Non-Inferiority — Non-inferiority p-value is calculated corresponding to the non-inferiority margin 0.1 unit; p = 0.0017, Repeated measures analysis; Change from baseline = Treatment + baseline EMSCI score + BR a/s MDI + stratification factor (prior treatment) + region + TI + treatment by TI; Least Square Mean Difference = 0.034, 95% CI 2-sided [-0.011 to 0.078], Standard Error of Mean 0.023 — [estimate comment as in outcome 1, analysis 1]

7. Other Pre Specified Outcome: Mean Change From Baseline in Night-Time Symptoms of COPD Instrument (NiSCI) Over 24 Weeks
Description: Change from baseline in the 6-item NiSCI Symptom Severity Score was derived by averaging the responses from a participant on the 6 item-level symptom scores (scored on a 4-point scale from 1 to 4, whereas 1= mild and 4= very severe). The NiSCI collected data about the frequency and severity of night-time symptoms and the impact of COPD symptoms on night-time awakenings in participants with COPD. Participants completed a daily ePRO questionnaire for their COPD symptoms. Baseline is defined as the average of the non-missing values from the ePRO data collected in the last 7 days before the randomization (Day 1).
Time Frame: From Baseline (Day -7) up to 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Glycopyrronium/Formoterol Fumarate | Umeclidinium/Vilanterol
Number analyzed (Participants) | 506 | 510
Units on a scale | -0.165 (0.019) | -0.207 (0.019)
Statistical Analysis 1: Comparison: Glycopyrronium/Formoterol Fumarate vs Umeclidinium/Vilanterol; Test type: Non-Inferiority — Non-inferiority p-value is calculated corresponding to the non-inferiority margin 0.1 unit; p = 0.0088, Repeated measures analysis; Change from baseline = Treatment + baseline NiSCI score + BR a/s MDI + stratification factor (prior treatment) + region + TI + treatment by TI; Least Square Mean Difference = 0.042, 95% CI 2-sided [-0.005 to 0.090], Standard Error of Mean 0.024 — [estimate comment as in outcome 1, analysis 1]

8. Other Pre Specified Outcome: Mean Change From Baseline in Daily Rescue (Albuterol/Salbutamol MDI) Use Over 24 Weeks
Description: The number of inhalations of rescue albuterol/salbutamol MDI was recorded in the participant ePRO in the morning and evening. Baseline is defined as the average of the non-missing values from the ePRO data collected in the last 7 days before the randomization (Day 1). a/s = albuterol/salbutamol.
Time Frame: From Baseline (Day -7) up to 24 weeks
Population: The rescue medication user analysis set included all participants in the FAS with average baseline rescue albuterol/salbutamol MDI use of >=1 inhalation/day. Only participants with data available for analysis are presented.
Measure: Least Squares Mean (Standard Error); unit: puffs/day
Arm/Group | Glycopyrronium/Formoterol Fumarate | Umeclidinium/Vilanterol
Number analyzed (Participants) | 456 | 454
puffs/day | -1.70 (0.16) | -2.35 (0.16)
Statistical Analysis 1: Comparison: Glycopyrronium/Formoterol Fumarate vs Umeclidinium/Vilanterol; Test type: Superiority; p = 0.9995, Repeated measures analysis; Change from baseline =Treatment + baseline rescue a/s MDI use + BR a/s MDI + stratification factor (prior treatment) + region + TI + treatment by TI; Least Square Mean Difference = 0.65, 95% CI 2-sided [0.26 to 1.04], Standard Error of Mean 0.20 — [estimate comment as in outcome 1, analysis 1]

9. Other Pre Specified Outcome: Mean Change From Baseline in COPD Assessment Test (CAT) Score Over 24 Weeks
Description: The CAT is used to quantify the impact of COPD symptoms on health status. The CAT has a scoring range of 0-40, and it is calculated as the sum of the responses given for each of the 8 items (scored on a 6-point scale from 0 to 5), with higher scores indicating a higher impact of COPD symptoms on health status. If the response to 1 of the 8 items is missing, the missing item was considered equal to the average of the 7 non-missing items for that participant. If more than 1 item is missing the score was considered missing. Baseline is defined as the latest assessment within 7 days before or at randomization (Day 1).
Time Frame: From Baseline (Day -7 or 1) up to 24 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Glycopyrronium/Formoterol Fumarate | Umeclidinium/Vilanterol
Number analyzed (Participants) | 506 | 510
Units on a scale | -2.97 (0.21) | -3.56 (0.22)
Statistical Analysis 1: Comparison: Glycopyrronium/Formoterol Fumarate vs Umeclidinium/Vilanterol; Test type: Non-Inferiority — Non-inferiority p-value is calculated corresponding to the non-inferiority margin 2.0 unit; p < 0.0001, Repeated measures analysis; Change from baseline = Treatment + baseline CAT score + BR a/s MDI + stratification factor (prior treatment) + region + visit + treatment by visit; Least Square Mean Difference = 0.59, 95% CI 2-sided [0.07 to 1.11], Standard Error of Mean 0.27 — [estimate comment as in outcome 1, analysis 1]

10. Primary Outcome: Mean Peak Change From Baseline in FEV1 Within 2 Hours Post-dosing Over 24 Weeks in FAS Population
Description: To assess the effects of GFF relative to UV on lung function in FAS population as measured by peak change from baseline in FEV1 is defined as the maximum of the FEV1 assessments within the 2 hours post-dosing time windows at each visit minus baseline using spirometry. Baseline is defined as the mean of the non-missing -60 and -30 minute values obtained prior to dosing at randomization (Day 1).
Time Frame: From Baseline (Day 1) up to 24 weeks
Population: The FAS included all randomized participants who received at least 1 inhalation of IP from the GFF or UV inhaler (active or placebo).
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Glycopyrronium/Formoterol Fumarate | Umeclidinium/Vilanterol
Number analyzed (Participants) | 552 | 552
mL | 299.1 (9.9) | 300.8 (9.9)
Statistical Analysis 1: Comparison: Glycopyrronium/Formoterol Fumarate vs Umeclidinium/Vilanterol; Test type: Superiority; p = 0.5516, Repeated measures analysis; [statistical method as in outcome 1, analysis 1]; Least Square Mean Difference = -1.7, 97.5% CI 2-sided [-30.3 to 27.0], Standard Error of Mean 12.8 — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: From Baseline (Day 1) up to 14 days after last IP dose, approximately 26 weeks.
Description: The safety analysis set included all participants who received at least 1 inhalation of the randomized active IP that they were assigned.
Arm/Group | Glycopyrronium/Formoterol Fumarate | Umeclidinium/Vilanterol
All-Cause Mortality (participants affected / at risk) | 3/552 | 3/552
Serious Adverse Events (participants affected / at risk) | 32/552 | 40/552
Other Adverse Events (participants affected / at risk) | 129/552 | 153/552
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glycopyrronium/Formoterol Fumarate (N=552) | Umeclidinium/Vilanterol (N=552)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 2 (2)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 1 (1)
Incarcerated hernia (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 16 (17) | 10 (12)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Essential hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Malignant hypertension (Vascular disorders) | 1 (1) | 0 (0)
Post thrombotic syndrome (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glycopyrronium/Formoterol Fumarate (N=552) | Umeclidinium/Vilanterol (N=552)
Vertigo (Ear and labyrinth disorders) | 5 (6) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 7 (8)
Constipation (Gastrointestinal disorders) | 1 (1) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 7 (8) | 13 (15)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 6 (6)
Toothache (Gastrointestinal disorders) | 1 (1) | 6 (6)
Nasopharyngitis (Infections and infestations) | 30 (32) | 36 (42)
Sinusitis (Infections and infestations) | 4 (4) | 6 (8)
Upper respiratory tract infection (Infections and infestations) | 10 (13) | 10 (13)
Viral upper respiratory tract infection (Infections and infestations) | 17 (18) | 26 (27)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (13) | 9 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (7)
Headache (Nervous system disorders) | 34 (52) | 41 (55)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 20 (22) | 20 (22)
Hypertension (Vascular disorders) | 13 (16) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-07-14): https://cdn.clinicaltrials.gov/large-docs/55/NCT03162055/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/55/NCT03162055/SAP_001.pdf